CLINICAL TRIAL: NCT05298072
Title: Identification of Novel Inflammation-related Biomarkers for Early Detection of Anthracycline-induced Cardiotoxicity in Breast Cancer Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Essen (Other)
Responsible Party: Sponsor
Other Study IDs: 22-10590-BO
Record Dates: First submitted 2022-03-17; First posted 2022-03-28 (Actual); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Cardiotoxicity; Breast Cancer; Heart Failure
MeSH Terms: conditions — Cardiotoxicity; Breast Neoplasms; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to identify possible set of inflammatory biomarkers before, during and after anthracycline-based chemotherapy in breast cancer patients to identify (sub)clinical chemotherapy-related cardiac dysfunctionCRCD to identify patients who would benefit from additional cardioprotective therapy.

ELIGIBILITY:
Inclusion Criteria:

* initial diagnosis of breast cancer
* planned Anthracycline-based therapy
* first-line chemotherapy
* first visit before initiation of chemotherapy

Exclusion Criteria:

* previous chemotherapy
* medical history of cardiac disease
* inflammation-modulating medication
* medication with RAS inhibitors
* pregnancy
* autoimmune disease
* drug addictions
* unwilling or unable to provide informed consent

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: all patients presenting to cardio-oncology unit complying with eligibility criteria
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2022-04 (Estimated); Primary Completion 2023-04 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Cardiotoxicity during observational period | continuous evaluation during observational period of 12 months
  Defined according to IC-OS 2021 Consensus Criteria